CLINICAL TRIAL: NCT05525013
Title: Effect of Simvastatin Versus Calcium Hydroxide Used as Intracanal Medicaments on Post-operative Pain and Total Amount of IL-6 and IL-8 in Periapical Fluids in Patients With Symptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Effect of Simvastatin Versus Calcium Hydroxide Intracanal Medications on Post-operative Pain and Interleukin 6 and 8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Essam Othman Ibrahim, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2022-8-30
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Periapical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: A Computerized random sequence will be generated using computer software (http://www.random.org/). The sequence generation will be done for the patients' numbers which results in a sequence of random numbers divided in two columns (A & B), where one column assigned for the intervention groups and one for the control group and kept with the co- supervisor. The patients will be allocated into either of the two groups with allocation ratio 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: After the participant is confirmed eligible for the study, the participant will drag an envelope and will be given a number. Based on this number the patient will be allocated to either intervention or control group after contacting the co- supervisor to reveal the assigned group of the current patient according to the generated random sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin as an intracanal medication
  Interventions: Drug: Simvastatin Powder
- Calcium hydroxide (Active Comparator): Calcium hydroxide intracanal medication
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Simvastatin Powder — Simvastatin gel placed as an intracanal medication
  Arms: Simvastatin
Drug: Calcium Hydroxide — Calcium hydroxide intracanal medication
  Arms: Calcium hydroxide

SUMMARY:
Comparing the effect of Simvastatin versus calcium hydroxide used as an intracanal medicament on Post-operative Pain and Total amount of IL-6 and IL-8 in Periapical Fluids of lower premolars in patients with Symptomatic Apical Periodontitis:

DETAILED DESCRIPTION:
Lower premolars with symptomatic apical periodontitis will be selected according to the eligibility and exclusion criteria and patients are then randomized to receive treatment either using simvastatin or calcium hydroxide intracanal medication for 1 week. The endodontic treatment will be completed in two visits. Postoperative pain will be assessed using the Numerical Rating scale at 6, 12, 24, 48 hours post-instrumentation and at 6, 12, 24, 48 hours post-obturation. Periapical fluid sample will be collected immediately post-instrumentation and 1 week later pre-obturation. The periapical samples will be analyzed for total amounts of IL-6 and IL-8.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Lower single rooted premolars:

  * Presence of pain with percussion.
  * Widening in the periodontal membrane space or with small sized periapical radiolucency.
  * Diagnosed clinically with symptomatic apical periodontitis.
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

* Medically compromised patients
* Pregnant women
* Patients who are allergic to non-steroidal anti-inflammatory drugs.
* Patients with two or more adjacent teeth requiring root canal therapy
* If analgesics or antibiotics have been administrated by the patient during the past two weeks preoperatively.
* Patients reporting bruxism or clenching.
* Teeth associated with acute periapical abscess, swelling or a fistulous tract.
* Greater than grade I mobility or pocket depth greater than 5mm.
* Non restorable teeth.
* Immature teeth.
* Teeth with previous endodontic treatment.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain incidence and intensity assessed with numerical rating scale | 6,12,24 and 48 hours post-instrumentation and 6,12,24 and 48 hours post-obturation
  0 (none) to 10 (severe) Numerical Pain Rating Scale

SECONDARY OUTCOMES:
Total amount of IL-6 and IL-8 in periapical fluids | Immediately post-instrumentation and pre-obturation (1 week post- instrumentation)
  Absorbance using ELISA test in Pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AA, Sun X, Hargreaves KM. Effect of calcium hydroxide on proinflammatory cytokines and neuropeptides. J Endod. 2008 Nov;34(11):1360-1363. doi: 10.1016/j.joen.2008.08.020. Epub 2008 Sep 17. PMID 18928847
- [Background] Sharma A, Sanjeev K, Selvanathan VMJ, Sekar M, Harikrishnan N. The evaluation of cytotoxicity and cytokine IL-6 production of root canal sealers with and without the incorporation of simvastatin: an invitro study. BMC Oral Health. 2022 Jan 11;22(1):6. doi: 10.1186/s12903-022-02039-y. PMID 35012572